CLINICAL TRIAL: NCT01129206
Title: Phase II Study of Pralatrexate and Docetaxel in Patients With Advanced Esophageal and Gastroesophageal Carcinoma Who Have Failed Prior Platinum-based Therapy.
Brief Title: Pralatrexate and Docetaxel in Treating Patients With Stage IV Esophageal or Gastroesophageal Cancer Who Have Failed Platinum-Based Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10018; NCI-2010-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinomas of the Gastroesophageal Junction; Recurrent Esophageal Cancer; Squamous Cell Carcinoma of the Esophagus; Stage IV Esophageal Cancer
Keywords: Gastroesophageal Cancer; Gastroesophageal Carcinoma; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma | interventions — 10-propargyl-10-deazaaminopterin; Docetaxel; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive pralatrexate IV over 3-5 minutes and docetaxel IV on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pralatrexate; Drug: docetaxel; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography

INTERVENTIONS:
Drug: pralatrexate — IVP(intravenous push)over 3-5 minutes on day 1 at a dose of 120 mg/m2.
  Other Names: FOLOTYN; PDX
Drug: docetaxel — Given Intravenous Piggyback (IVPB)as one-hour infusion at a dose of 3 mg/m2 on day 1 of a cycle. cycle defined as 14 days.
  Other Names: RP 56976; Taxotere; TXT
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; fluorodeoxyglucose F 18
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
RATIONALE: Pralatrexate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pralatrexate together with docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pralatrexate together with docetaxel works in treating patients with stage IV esophageal or gastroesophageal cancer who have failed platinum-based therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall response rate CR & PR(Complete Response + Partial Response)as assessed by RECIST (Response Evaluation Criteria in Solid Tumors v 1.1) of the combination of pralatrexate and docetaxel in patients with advanced esophageal and gastroesophageal carcinomas.

SECONDARY OBJECTIVES:

I. Evaluation of progression free survival and overall survival. II. Correlation of FDG(fludeoxyglucose)PET(positron emission tomography)response defined as a 35% reduction in SUV(standard uptake value)during the early course of chemotherapy to progression free and overall survival in addition to radiographic response as measured by RECIST v 1.1 criteria on CT imaging.

OUTLINE:

Patients receive pralatrexate IV over 3-5 minutes and docetaxel IV on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion

* Pathologically confirmed unresectable advanced or metastatic carcinoma of the esophagus or gastroesophageal junction
* Established histological confirmation of squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction
* Stage IV disease
* Must have received platinum-based therapy; this includes definitive, adjuvant and metastatic treatments
* No more than 3 chemotherapeutic treatment regimens permitted; this includes concurrent chemoradiation
* Radiation therapy allowed if > 4 weeks have elapsed
* Must be off therapy for 4 weeks prior to enrollment
* Measurable disease as defined by RECIST v 1.1 criteria
* ECOG (Eastern Cooperative Oncology Group)PS(Performance status)of 0 to 2
* Predicted life expectancy of at least 12 weeks
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial and for three months after completion of treatment
* Marrow: ANC(absolute neutrophil count)> 1,000/mm^3
* Marrow: Hemoglobin > 9.0 g/dl
* Marrow: Platelet Count > 100,000/mm^3
* Renal: Serum creatinine =< 1.5 g/dL
* Hepatic: Serum bilirubin < 1.5 x ULN(upper limit of normal) and AST (aspartate aminotransferase) and ALT (Alanine aminotransferase)=< 2.5 x ULN
* Prior minor surgeries (such as laparoscopies) must have occurred at least 14 days prior to study enrollment; prior minor procedures such as biopsies and mediport placement must have occurred at least 48 hours prior to study enrollment
* All patients must have signed an informed consent indicating that they are aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts
* History of allergic reactions attributed to compounds of similar chemical composition to agents used in the study

Exclusion

* Pregnant or lactating women
* Patients with any severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for study entry
* Any malignant condition for which one has received treatment in the last two years excluding squamous or basal cell carcinomas
* Patients with untreated brain metastases
* Patients must not have grade 2 or higher baseline peripheral neuropathy, according to CTCAE v 4.0
* Patients must have NO continuing acute toxic effects (except alopecia) of any prior radiotherapy, chemotherapy, or surgical procedures; all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE v 4.0) Grade =< 1 prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Saab, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Petullo B, Wei L, Yereb M, Neal A, Rose J, Bekaii-Saab T, Wu C. A phase II study of biweekly pralatrexate and docetaxel in patients with advanced esophageal and gastroesophageal carcinoma that have failed first-line platinum-based therapy. J Gastrointest Oncol. 2015 Jun;6(3):336-40. doi: 10.3978/j.issn.2078-6891.2015.011. PMID 26029462
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II single-arm, open label trial performed at The Ohio State University James Cancer Hospital.
Groups:
- Arm I: Pralatrexate and Docetaxel: Patients receive pralatrexate IV over 3-5 minutes and docetaxel IV on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  pralatrexate: IVP(intravenous push)over 3-5 minutes on day 1 at a dose of 120 mg/m2.
  docetaxel: Given Intravenous Piggyback (IVPB)as one-hour infusion at a dose of 3 mg/m2 on day 1 of a cycle. cycle defined as 14 days.
  fludeoxyglucose F 18: Correlative studies
  positron emission tomography: Correlative studies
Period: Overall Study
Arm/Group | Arm I: Pralatrexate and Docetaxel
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 63.5 [55 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Approximately three years
Measure: Number; unit: patients
Arm/Group | Arm I: Pralatrexate and Docetaxel
Number analyzed (Participants) | 6
patients
  Stable disease | 2
  Progressive disease | 4

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Approximately three years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Pralatrexate and Docetaxel
Number analyzed (Participants) | 6
months | 1.9 [0.8 to 7.2]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was determined from the date of start of therapy to death frm any cause.
Time Frame: Approximately five years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 6
months | 5.5 [0.8 to 11.7]

4. Secondary Outcome: Correlation of FDG PET Response With Response Rate
Description: Radiological assessment of tumor response was performed by computed tomography (CT) and positron emission tomography (PET) every four cycles of therapy and responses were measured according to RECIST and PERCIST criteria.
Time Frame: Approximately three years
Population: 2 patients not evaluable for response applying the PERCIST criteria per PET
Measure: Number; unit: patients
Arm/Group | PERCIST Criteria Per PET | RECIST Criteria Per CT
Number analyzed (Participants) | 4 | 6
patients
  Progressive Disease | 0 | 4
  Stable Disease | 2 | 2
  Partial Response | 2 | 0

ADVERSE EVENTS:
Description: Toxicities were defined by the National Cancer Institutes CTCAE version 3.0
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=6)
Lymphopenia (Investigations) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Investigations) | 2 (2)
Mucocitis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes